CLINICAL TRIAL: NCT05594758
Title: Named Patient Program for Providing Access to Olverembatinib (HQP1351) to Countries Where the Drug is Not Available
Brief Title: Named Patient Program for Olverembatinib (HQP1351)
Status: Available | Type: Expanded Access
Sponsor: Ascentage Pharma Group Inc. (Industry)
Collaborators: Tanner Pharma Group (Other)
Responsible Party: Sponsor
Other Study IDs: NPP Olverembatinib
Record Dates: First submitted 2022-10-21; First posted 2022-10-26 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

Keywords: Named Patient Program
MeSH Terms: interventions — olverembatinib

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Olverembatinib — Oral Olverembatinib

SUMMARY:
This program will allow eligible patients access to Ascentage Pharma's novel drug candidate Olverembatinib (approved in China) on a named patient basis in over 100 countries ( with the exception of the USA and China) and regions where the drug is not available.

DETAILED DESCRIPTION:
Olverembatinib is a novel third generation BCR-ABL inhibitor that can effectively target a spectrum of BCR-ABL mutants, including the T315I mutation. Olverembatinib is approved in China for the treatment of adult patients with tyrosine kinase inhibitor (TKI)-resistant chronic phase chronic myeloid leukemia (CP-CML) or accelerated-phase CML (AP-CML) harboring the T315I mutation as confirmed by a validated diagnostic test1.

ELIGIBILITY:
Inclusion Criteria:

• Patients who are suitable to receive Olverembatinib and for whom there is reasonable expectation that Olverembatinib may provide clinical benefit based on the medical judgment of their prescribing physician.

Exclusion Criteria:

* Existing risks of serious Arterial occlusive events (AOE), including myocardial infarction, stroke, stenosis of large arterial vessels of the brain, severe peripheral vascular disease, and recent revascularization procedures
* Existing risks of serious Venous thromboembolic events (VTEs), including deep venous thrombosis, pulmonary embolism, and retinal vein thrombosis
* Existing serious heart conditions, including acute/chronic heart failure, coronary artery disease
* Existing conditions of severe liver malfunction
* Existing conditions of severe myelosuppression
* Existing conditions of severe hemorrhage
* Pregnant or baby feeding

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult